CLINICAL TRIAL: NCT00082914
Title: Phase II Evaluation of Denileukin Diftitox in Patients With Metastatic Melanoma or Metastatic Kidney Cancer
Brief Title: Denileukin Diftitox in Treating Patients With Metastatic Melanoma or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000361715; NCI-04-C-0134; NCT00078702 (obsolete NCT alias)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-12

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — denileukin diftitox

INTERVENTIONS:
Biological: denileukin diftitox

SUMMARY:
RATIONALE: Denileukin diftitox may be able to make the body build an immune response to kill tumor cells.

PURPOSE: This phase II trial is studying how well denileukin diftitox works in treating patients with metastatic melanoma or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical response in patients with metastatic melanoma or metastatic kidney cancer treated with denileukin diftitox.

Secondary

* Determine whether changes occur in levels of CD4-positive CD25-positive lymphocytes in the peripheral blood of these patients before and after treatment with this drug.
* Determine the toxicity profile of this drug in these patients.

OUTLINE: Patients are stratified according to disease type (metastatic melanoma vs metastatic kidney cancer).

Patients receive denileukin diftitox IV over 1 hour on days 1-5, 21-25, 42-46, and 63-67. Treatment repeats every 84 days (12 weeks) for up to a maximum total of 5 courses in the absence of disease progression, autoimmune ocular toxicity attributable to denileukin diftitox, or any other unacceptable toxicity. At any time during therapy, patients achieving a complete response receive 1 additional course of therapy after the complete response.

PROJECTED ACCRUAL: A total of 10-96 patients (5-48 per stratum) will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Melanoma
  * Kidney cancer
* Metastatic disease
* Measurable disease
* Documented disease progression while receiving standard therapy
* No resectable local or regional disease

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 90,000/mm^3
* Lymphocyte count ≥ 500/mm^3
* No concurrent coagulation disorders

Hepatic

* Bilirubin ≤ 2.0 mg/dL (< 3.0 mg/dL for patients with Gilbert's syndrome)
* AST and ALT < 3 times normal
* Albumin ≥ 2.5 g/dL
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine ≤ 2.0 mg/dL

Cardiovascular

* Normal thallium stress test*
* No prior myocardial infarction
* No history of severe coronary artery disease
* No major medical illness of the cardiovascular system NOTE: *For patients > 50 years of age OR who have a history of cardiovascular disease

Pulmonary

* No major medical illness of the respiratory system

Immunologic

* HIV negative
* No active systemic infection
* No presence of opportunistic infections
* No primary or secondary immunodeficiency
* No autoimmune disease
* No other known immunodeficiency

Other

* No sensitivity to denileukin diftitox or any of its components (e.g., diphtheria toxin, interleukin-2, or excipients)
* Willing to undergo leukapheresis
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior treatment with interleukin-2 allowed provided the patient's disease status required this therapy

Chemotherapy

* Recovered from prior chemotherapy

Endocrine therapy

* No concurrent systemic steroids

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* More than 3 weeks since prior systemic anticancer therapy
* No other concurrent systemic anticancer therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-03; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Clinical response

SECONDARY OUTCOMES:
Changes in levels of CD4-positive CD25-positive lymphocytes in the peripheral blood
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland